CLINICAL TRIAL: NCT07268950
Title: Structured Simulation-Based Training to Develop Laparoscopic and Thoracoscopic Skills in Thoracic Surgery and Rotating Surgical Residents: A Component-Based Educational Model
Brief Title: Structured Simulation Training for Laparoscopic and Thoracoscopic Skills in Thoracic Surgery Residents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Caner İşevi, MD, Principal Investigator, Ondokuz Mayıs University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: B.30.2.ODM.0.20.08/498
Record Dates: First submitted 2025-11-25; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Surgical Education; Simulation-based Training; Resident Training

STUDY DESIGN:
Intervention Model Description: Participants will receive a structured simulation-based training program consisting of standardized laparoscopic and thoracoscopic skill modules. All participants complete pre-training and post-training assessments using the same protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Structured Simulation Training (Experimental): Participants will undergo a standardized simulation-based training program designed to develop laparoscopic and thoracoscopic technical skills. Training includes camera navigation, tissue dissection, stapling, and suturing tasks performed on box trainers, artificial models, and bovine tissues in a controlled laboratory setting. All participants complete baseline (pre-training) and post-training evaluations using OSATS scoring, self-assessment surveys, and performance timing. No clinical procedures, live animals, or patient interactions occur during the study.
  Interventions: Behavioral: Structured Simulation-Based Surgical Training

INTERVENTIONS:
Behavioral: Structured Simulation-Based Surgical Training — Participants will complete a structured simulation-based training curriculum designed to improve fundamental laparoscopic and thoracoscopic surgical skills. The program includes standardized modules on camera navigation, tissue handling, dissection, stapling, and suturing, performed on box trainers, artificial models, and bovine tissues. Training occurs in a controlled laboratory environment with faculty supervision and predefined performance goals. No real patients, clinical procedures, or live animals are involved. All participants undergo pre- and post-training performance assessment using OSATS scoring, task completion time, and self-evaluation surveys.
  Other Names: Component-Based Laparoscopic-Thoracoscopic Training; Simulation Skills Curriculum

SUMMARY:
This study aims to improve basic laparoscopic and thoracoscopic skills in thoracic surgery residents and rotating surgical residents through a structured simulation-based training program. Participants will complete hands-on practice sessions using box trainers, artificial models, and bovine tissues in a controlled, non-patient setting.

Before and after the training, participants will complete self-assessment surveys and a standardized technical skills evaluation (OSATS). The study will compare these results to measure changes in technical performance, confidence, and learning needs. No real patients, live animals, or clinical procedures are involved, and there are no expected medical risks.

The goal of this study is to determine whether structured simulation training is effective, practical, and acceptable for surgical education, and whether it can support safer transition to real operating room experience in the future.

ELIGIBILITY:
Inclusion Criteria:

* Thoracic surgery residents OR rotating general surgery/cardiovascular surgery residents
* Age ≥18 years
* Actively enrolled in an accredited residency training program
* Willingness to participate in hands-on simulation training
* Ability to provide informed consent
* Able to complete video-recorded performance assessments

Exclusion Criteria:

* Prior advanced laparoscopic or thoracoscopic fellowship training
* Inability to safely handle surgical instruments (e.g., significant musculoskeletal limitation)
* Previous participation in a similar structured simulation program within the past 12 months
* Declines consent or withdraws participation
* Unable to attend required training and assessment sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in Total OSATS Score | Baseline (pre-training) and immediately after completion of the training program (within 1 week)
  Technical skill performance will be assessed using the Objective Structured Assessment of Technical Skills (OSATS), consisting of a global rating scale and task-specific checklist (total score range 0-35). Each participant will complete the same standardized tasks before and after the simulation training. The primary outcome is the within-subject change (post-training minus pre-training) in total OSATS score.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University Medical Faculty, Department of Thoracic Surgery, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the sample size is small and performance videos, OSATS scores, and survey results may allow indirect identification of surgical trainees. Data are collected solely for educational and research purposes within a single institution and will be stored securely according to ethics committee requirements. Only aggregated and de-identified results will be reported in publications and presentations.